CLINICAL TRIAL: NCT03340766
Title: A Phase 1b Open Label Study Investigating the Safety and Efficacy of Blinatumomab in Combination With Pembrolizumab in Adult Subjects With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Study Investigating the Safety and Efficacy of Blinatumomab in Combination With Pembrolizumab in Adults With Relapsed or Refractory Diffuse Large B Cell Lymphoma (DLBCL)
Acronym: HARBOUR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20150290; 2016-002191-27 (EudraCT Number); PN348 (Other: Merck Protocol Number)
Expanded Access: NCT02187354 (No longer available)
Record Dates: First submitted 2017-10-23; First posted 2017-11-14 (Actual); Results first posted 2022-02-25 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-07

CONDITIONS: Relapsed or Refractory Diffuse Large B Cell Lymphoma (DLBCL)
Keywords: DLBCL Relapsed post-autologous or allogeneic hematopoietic stem cell transplantation (HSCT); Antibodies; Bispecific in combination with PD-1/PD-L1 inhibitor
MeSH Terms: conditions — Recurrence; Lymphoma, Large B-Cell, Diffuse | interventions — blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort Ia: Blinatumomab 9/28 µg/day + Pembrolizumab (Experimental): Participants received blinatumomab administered as a continuous intravenous infusion (CIVI) for 8 weeks followed by a 28-day treatment-free interval. Participants with stable disease or better may have received a second 28-day consolidation cycle. The starting dose of each cycle was 9 µg/day for the first 7 days then 28 µg/day for the remaining days of treatment.
  Starting on Day 15 participants also received 200 mg pembrolizumab administered by intravenous (IV) infusion every 3 weeks (Q3W) until disease progression or for up to 35 cycles.
  Interventions: Drug: Blinatumomab; Drug: Pembrolizumab
- Cohort IIa: Blinatumomab 9/28/56 µg/day + Pembrolizumab (Experimental): Participants received blinatumomab administered as a continuous intravenous infusion for 8 weeks followed by a 28-day treatment-free interval. Participants with stable disease or better may have received a second 28-day consolidation cycle. The starting dose of each cycle was 9 µg/day for the first 7 days, 28 µg/day for 7 days then 56 µg/day for the remaining days of treatment.
  Starting on Day 19 participants also received 200 mg pembrolizumab administered by IV infusion Q3W until disease progression or for up to 35 cycles.
  Interventions: Drug: Blinatumomab; Drug: Pembrolizumab
- Cohort IIIa: Blinatumomab 9/28/112 µg/day + Pembrolizumab (Experimental): Participants received blinatumomab administered as a continuous intravenous infusion for 8 weeks followed by a 28-day treatment-free interval. Participants with stable disease or better may have received a second 28-day consolidation cycle. The starting dose of each cycle was 9 µg/day for the first 7 days, 28 µg/day for 7 days then 112 µg/day for the remaining days of treatment.
  Starting on Day 19 participants also received 200 mg pembrolizumab administered by IV infusion Q3W until disease progression or for up to 35 cycles.
  Interventions: Drug: Blinatumomab; Drug: Pembrolizumab
- Expansion Cohort (Experimental): This cohort will test the maximum tolerated dose of blinatumomab in combination with pembrolizumab identified in Part 1 of the study.
  Interventions: Drug: Blinatumomab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Blinatumomab — Up to 2 cycles of blinatumomab may be given, where cycle 1 lasts 8 weeks, and cycle 2 lasts 28 days. The treatment is given as a continuous intravenous infusion.
  Other Names: Blincyto; AMG 103; Formerly known as MT103 or bscCD19xCD3
Drug: Pembrolizumab — One cycle of pembrolizumab is a 200 mg IV injection lasting 30 minutes. One cycle will be given every 3 weeks until disease progression, or for a maximum of 35 cycles.
  Other Names: Keytruda; MK-3475

SUMMARY:
The primary objective of the study is to determine the maximum tolerated dose (MTD) of blinatumomab in combination with pembrolizumab in adults with relapsed or refractory (r/r) DLBCL.

DETAILED DESCRIPTION:
The study was planned as 2 parts:

* Part 1 will test the safety of up to 3 different blinatumomab target dose levels in combination with pembrolizumab in a rolling 6 design. A Dose Level Review Team (DLRT) will review the safety data to evaluate possible drug effects and dose-limiting toxicities (DLTs).
* Part 2 will consist of an expansion cohort to assess pharmacokinetics (PK), safety, and preliminary efficacy data at the chosen target dose. The part 2 dose will be determined by the totality of the clinical data from part 1 as determined by the DLRT.

Based on the results from Part 1, a decision was made not to proceed with Part 2 of this study.

Secondary objectives of the study are to evaluate the safety, efficacy, and pharmacokinetics (PK) of blinatumomab in combination with pembrolizumab. Tumor response will be evaluated according to the Revised Response Criteria for Malignant Lymphoma (Cheson et al, 2007). With implementation of Protocol Amendment 5, response will also be assessed according to the Lugano Classification (Cheson et al, 2014). Only participants enrolled after implementation of Protocol Amendment 5 (03 December 2019) will have tumor assessments using the Lugano criteria.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed diffuse large B-cell lymphoma that is either:
* Refractory after at least one regimen of systemic chemotherapy and/or targeted therapy, or
* In first or later relapse if have received at least 2 systemic regimens since time of diagnosis, or
* Relapsed post-autologous or allogeneic hematopoietic stem cell transplantation (HSCT) with adequate organ function after proximity to transplantation time exclusions
* Have measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Life expectancy of ≥ 12 weeks in the opinion of the Investigator
* Biopsy proven DLBCL (biopsy proven at least at primary diagnosis of DLBCL)

Other Inclusion Criteria May Apply

Exclusion Criteria:

* Richter's transformation (DLBCL arising in the setting of prior chronic lymphocytic leukemia) or primary mediastinal B cell lymphoma (PMBCL)
* History or presence of clinically relevant central nervous system pathology such as epilepsy, paresis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.
* Has a diagnosis of immunodeficiency or has received systemic steroid therapy (in excess of 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of protocol specified therapy.
* Has undergone prior allogeneic HSCT:
* within the last 5 years OR
* greater than 5 years ago but has active graft versus host disease (GvHD) requiring systemic treatment.
* Has received autologous HSCT within 6 weeks prior to start of treatment.

Other Exclusion Criteria May Apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2023-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (22):
- United States (3):
  - Research Site, La Jolla, California
  - Research Site, Charleston, South Carolina
  - Research Site, Greenville, South Carolina
- Australia (7):
  - Research Site, Darlinghurst, New South Wales
  - Research Site, St Leonards, New South Wales
  - Research Site, Adelaide, South Australia
  - Research Site, East Melbourne, Victoria
  - Research Site, Geelong, Victoria
  - Research Site, Melbourne, Victoria
  - Research Site, Murdoch, Western Australia
- France (3):
  - Research Site, Créteil
  - Research Site, Nantes
  - Research Site, Pierre-Bénite
- Germany (3):
  - Research Site, Heidelberg
  - Research Site, Ulm
  - Research Site, Würzburg
- Netherlands (2):
  - Research Site, Maastricht
  - Research Site, Rotterdam
- Spain (4):
  - Research Site, Santander, Cantabria
  - Research Site, Salamanca, Castille and León
  - Research Site, Barcelona, Catalonia
  - Research Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 11 centers in Australia, France, Netherlands, Spain, and the United States.
  The study was planned as 2 parts. Based on the results from Part 1, a decision was made not to proceed with Part 2 of the study.
Pre-assignment Details: Participants were enrolled into each dose cohort sequentially using a rolling 6 study design. A Dose Level Review Team (DLRT) reviewed the safety data to evaluate possible drug effects and dose-limiting toxicities (DLTs).
Groups:
- Cohort Ia: Blinatumomab 9/28 µg/Day + Pembrolizumab: Participants in Cohort Ia received blinatumomab administered as a continuous intravenous infusion (CIVI) for 8 weeks followed by a 28-day treatment-free interval. Participants with stable disease or better may have received a second 28-day consolidation cycle. The starting dose of each cycle was 9 µg/day for the first 7 days, then 28 µg/day for the remaining 21 days of treatment. Starting on study Day 15 participants also received 200 mg pembrolizumab administered by IV infusion every 3 weeks (Q3W) until disease progression or for up to 35 cycles.
- Cohort IIa: Blinatumomab 9/28/56 µg/Day + Pembrolizumab: Participants in Cohort IIa received blinatumomab administered as a CIVI for 8 weeks followed by a 28-day treatment-free interval. Participants with stable disease or better may have received an additional 28-day consolidation cycle. The starting dose of each cycle was 9 µg/day for the first 7 days, 28 µg/day for 7 days, then 56 µg/day for the remaining 21 days of treatment. Starting on study Day 19 participants also received 200 mg pembrolizumab administered by IV infusion Q3W until disease progression or for up to 35 cycles.
- Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab: Participants in Cohort IIIa received blinatumomab administered as a CIVI for 8 weeks followed by a 28-day treatment-free interval. Participants with stable disease or better may have received an additional 28-day consolidation cycle. The starting dose of each cycle was 9 µg/day for the first 7 days, 28 µg/day for 7 days, then 112 µg/day for the remaining 21 days of treatment. Starting on study Day 19 participants also received 200 mg pembrolizumab administered by IV infusion Q3W until disease progression or for up to 35 cycles.
Period: Overall Study
Arm/Group | Cohort Ia: Blinatumomab 9/28 µg/Day + Pembrolizumab | Cohort IIa: Blinatumomab 9/28/56 µg/Day + Pembrolizumab | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab
Started | 12 | 10 | 9
Received Blinatumomab | 12 | 10 | 9
Received Pembrolizumab | 10 | 7 | 7
Completed | 4 | 2 | 1
Not Completed | 8 | 8 | 8
Not completed — Withdrawal by Subject | 2 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Death | 6 | 7 | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: Included all participants who received blinatumomab.
Groups:
- Cohort Ia: Blinatumomab 9/28 µg/Day + Pembrolizumab: Participants in Cohort Ia received blinatumomab administered as CIVI for 8 weeks followed by a 28-day treatment-free interval. Participants with stable disease or better may have received a second 28-day consolidation cycle. The starting dose of each cycle was 9 µg/day for the first 7 days, then 28 µg/day for the remaining 21 days of treatment. Starting on study Day 15 participants also received 200 mg pembrolizumab administered by IV infusion Q3W until disease progression or for up to 35 cycles.
- Total: Total of all reporting groups
Arm/Group | Cohort Ia: Blinatumomab 9/28 µg/Day + Pembrolizumab | Cohort IIa: Blinatumomab 9/28/56 µg/Day + Pembrolizumab | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab | Total
Number analyzed (Participants) | 12 | 10 | 9 | 31
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 7 | 3 | 4 | 14
  From 65-84 years | 5 | 7 | 5 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 5 | 9
  Male | 10 | 8 | 4 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 9 | 8 | 29
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 0 | 2
  White | 11 | 7 | 8 | 26
  Other | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Dose-limiting toxicities were grade 3-5 adverse events that occurred during the DLT-evaluation period that were judged by the Investigator to be possibly, probably or definitely related to study drug administration.
  All toxicities were graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0:
  * Grade 3: Severe or medically significant but not immediately life-threatening.
  * Grade 4: Life-threatening.
  * Grade 5: Death.
Time Frame: The DLT evaluation period was 42 days from initiation of pembrolizumab treatment (Day 15 for Cohort Ia and Day 19 for Cohorts IIa and IIIa)
Population: DLT Analysis Set: Included participants who experienced a DLT, OR were removed from treatment for an adverse event/toxicity that was not a DLT or for other reasons and had been exposed to study treatment for ≥ 12 days OR completed the DLT evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort Ia: Blinatumomab 9/28 µg/Day + Pembrolizumab | Cohort IIa: Blinatumomab 9/28/56 µg/Day + Pembrolizumab | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab
Number analyzed (Participants) | 10 | 6 | 5
Participants | 1 | 0 | 2

2. Secondary Outcome: Objective Response Rate During the First 12 Weeks Using Revised Response Cheson Criteria
Description: Objective response rate is defined as the percentage of participants with either a complete response (CR) or a partial response (PR):
  * CR: Disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy: If fluorodeoxyglucose (FDG)-avid or positron emission tomography (PET) positive before therapy, a residual mass of any size is permitted if it is PET negative; For variably FDG-avid or if a pretreatment PET scan was negative, all lymph nodes and nodal masses must have regressed on computed tomography (CT) to normal size. Spleen or liver should not be palpable and normal size. Bone marrow infiltrate must have cleared or be negative by immunohistochemistry.
  * PR: Regression of measurable disease and no new sites (≥ 50% decrease in size of up to six of the largest dominant nodes or nodal masses and splenic and hepatic nodules).
  Participants with no post-baseline response assessments were considered non-responders.
Time Frame: First 12 weeks of blinatumomab treatment
Population: Full Analysis Set: Included all participants who received blinatumomab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort Ia: Blinatumomab 9/28 µg/Day + Pembrolizumab | Cohort IIa: Blinatumomab 9/28/56 µg/Day + Pembrolizumab | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab
Number analyzed (Participants) | 12 | 10 | 9
percentage of participants | 16.7 (2.1) [2.1 to 48.4] | 30.0 (6.7) [6.7 to 65.3] | 33.3 (7.5) [7.5 to 70.1]

3. Secondary Outcome: Cohort IIIa Only: Objective Response Rate During the First 12 Weeks Using the Lugano Classification
Description: Objective response rate is defined as the percentage of participants with either a complete metabolic response (CMR) or a partial metabolic response (PMR):
  * CMR: For PET-CT-based response, score of 1-3 on the Deauville five-point scale (5PS) for lymph nodes and extralymphatic sites, no evidence of FDG-avid disease in marrow. For CT-based response, target nodes/masses regress to 1.5 cm in longest transverse diameter, no extralymphatic sites of disease, normal bone marrow morphology
  * PMR: For PET-CT-based response, score of 4 or 5 on 5PS with reduced uptake compared to baseline for lymph nodes and extralymphatic sites, residual uptake reduced compared to baseline in the bone marrow. For CT-based response, ≥ 50% decrease in sum of the product of the perpendicular diameters of up to 6 target measurable nodes and extranodal sites, spleen must have regressed by > 50% in length beyond normal.
  Participants with no post-baseline response assessments were considered non-responders.
Time Frame: First 12 weeks of blinatumomab treatment
Population: Full Analysis Set: Included all participants who received blinatumomab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab
Number analyzed (Participants) | 9
percentage of participants | 11.1 (0.3) [0.3 to 48.3]

4. Secondary Outcome: Objective Response Rate During the Treatment Period Using Revised Response Cheson Criteria
Description: Objective response rate is defined as the percentage of participants with either a CR or a PR according to the Revised Response Criteria (2007):
  * CR: Disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy: If FDG-avid or PET positive before therapy, a residual mass of any size is permitted if it is PET negative; For variably FDG-avid or if a pretreatment PET scan was negative, all lymph nodes and nodal masses must have regressed on CT to normal size. Spleen or liver should not be palpable and normal size. Bone marrow infiltrate must have cleared or be negative by immunohistochemistry.
  * PR: Regression of measurable disease and no new sites (≥ 50% decrease in size of up to six of the largest dominant nodes or nodal masses and splenic and hepatic nodules).
  Participants with no post-baseline response assessments were considered non-responders.
Time Frame: From Day 1 to 30 days after last dose of either blinatumomab or pembrolizumab administration; the overall median duration of treatment was 87 days.
Population: Full Analysis Set: Included all participants who received blinatumomab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort Ia: Blinatumomab 9/28 µg/Day + Pembrolizumab | Cohort IIa: Blinatumomab 9/28/56 µg/Day + Pembrolizumab | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab
Number analyzed (Participants) | 12 | 10 | 9
percentage of participants | 25.0 (5.5) [5.5 to 57.2] | 40.0 (12.2) [12.2 to 73.8] | 33.3 (7.5) [7.5 to 70.1]

5. Secondary Outcome: Cohort IIIa Only: Objective Response Rate During the Treatment Period Using the Lugano Classification
Description: Objective response rate is defined as the percentage of participants with either a CMR or a CMR.
  * CMR: For PET-CT-based response, score of 1-3 on the Deauville 5PS for lymph nodes and extralymphatic sites, no evidence of FDG-avid disease in marrow. For CT-based response, target nodes/masses regress to 1.5 cm in longest transverse diameter, no extralymphatic sites of disease, normal bone marrow morphology
  * PMR: For PET-CT-based response, score of 4 or 5 on 5PS with reduced uptake compared to baseline for lymph nodes and extralymphatic sites, residual uptake reduced compared to baseline in the bone marrow. For CT-based response, ≥ 50% decrease in sum of the product of the perpendicular diameters of up to 6 target measurable nodes and extranodal sites, spleen must have regressed by > 50% in length beyond normal.
  Participants with no post-baseline response assessments were considered non-responders.
Time Frame: From study Day 1 to 30 days after last dose of either blinatumomab or pembrolizumab administration; the overall median duration of treatment was 87 days.
Population: Full Analysis Set: Included all participants who received blinatumomab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab
Number analyzed (Participants) | 9
percentage of participants | 11.1 (0.3) [0.3 to 48.3]

6. Secondary Outcome: Complete Response Rate During the First 12 Weeks Using the Revised Response Cheson Criteria
Description: Complete response rate is defined as the percentage of participants with a CR according to the Revised Response Criteria (2007):
  - CR: Disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy: If FDG-avid or PET positive before therapy, a residual mass of any size is permitted if it is PET negative; For variably FDG-avid or if a pretreatment PET scan was negative, all lymph nodes and nodal masses must have regressed on CT to normal size. Spleen or liver should not be palpable and normal size. Bone marrow infiltrate must have cleared or be negative by immunohistochemistry.
  Participants with no post-baseline response assessments were considered non-responders.
Time Frame: First 12 weeks of blinatumomab treatment
Population: Full Analysis Set: Included all participants who received blinatumomab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort Ia: Blinatumomab 9/28 µg/Day + Pembrolizumab | Cohort IIa: Blinatumomab 9/28/56 µg/Day + Pembrolizumab | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab
Number analyzed (Participants) | 12 | 10 | 9
percentage of participants | 0.0 (0.0) [0.0 to 26.5] | 20.0 (2.5) [2.5 to 55.6] | 11.1 (0.3) [0.3 to 48.3]

7. Secondary Outcome: Cohort IIIa Only: Complete Response Rate During the First 12 Weeks Using the Lugano Classification
Description: Complete response rate is defined as the percentage of participants with a CMR according to the Lugano classification (2014):
  CMR: For PET-CT-based response, score of 1-3 on the Deauville 5PS for lymph nodes and extralymphatic sites, no evidence of FDG-avid disease in marrow. For CT-based response, target nodes/masses regress to 1.5 cm in longest transverse diameter, no extralymphatic sites of disease, normal bone marrow morphology.
  Participants with no post-baseline response assessments were considered non-responders.
Time Frame: First 12 weeks of blinatumomab treatment
Population: Full Analysis Set: Included all participants who received blinatumomab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab
Number analyzed (Participants) | 9
percentage of participants | 11.1 (0.3) [0.3 to 48.3]

8. Secondary Outcome: Complete Response Rate During the Treatment Period Using the Revised Response Cheson Criteria
Description: Complete response rate is defined as the percentage of participants with a complete response according to the Revised Response Criteria (2007):
  - CR: Disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy: If FDG-avid or PET positive before therapy, a residual mass of any size is permitted if it is PET negative; For variably FDG-avid or if a pretreatment PET scan was negative, all lymph nodes and nodal masses must have regressed on CT to normal size. Spleen or liver should not be palpable and normal size. Bone marrow infiltrate must have cleared or be negative by immunohistochemistry.
  Participants with no post-baseline response assessments were considered non-responders.
Time Frame: as for outcome 4
Population: Full Analysis Set: Included all participants who received blinatumomab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort Ia: Blinatumomab 9/28 µg/Day + Pembrolizumab | Cohort IIa: Blinatumomab 9/28/56 µg/Day + Pembrolizumab | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab
Number analyzed (Participants) | 12 | 10 | 9
percentage of participants | 16.7 (2.1) [2.1 to 48.4] | 30.0 (6.7) [6.7 to 65.3] | 11.1 (0.3) [0.3 to 48.3]

9. Secondary Outcome: Cohort IIIa Only: Complete Response Rate During the Treatment Period Using the Lugano Classification
Description: Complete response rate is defined as the percentage of participants with a CMR according to the Lugano classification (2014):
  - CMR: For PET-CT-based response, score of 1-3 on the Deauville 5PS for lymph nodes and extralymphatic sites, no evidence of FDG-avid disease in marrow. For CT-based response, target nodes/masses regress to 1.5 cm in longest transverse diameter, no extralymphatic sites of disease, normal bone marrow morphology.
  Participants with no post-baseline response assessments were considered non-responders.
Time Frame: as for outcome 4
Population: Full Analysis Set: Included all participants who received blinatumomab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab
Number analyzed (Participants) | 9
percentage of participants | 11.1 (0.3) [0.3 to 48.3]

10. Secondary Outcome: Progression Free Survival by the Revised Response Cheson Criteria
Description: Progression-free survival was calculated as the time from the date of the first dose of blinatumomab until the date of diagnosis of progression of lymphoma using the Cheson revised response criteria (2007), or date of death, whichever was earliest.
  Participants who were alive and did not have progression were censored at the last radiological non-missing evaluable tumor assessment date.
  Progressive disease per the revised response criteria is any new lesion or increase of 50% or greater in size of nodal masses or lesions or new or recurrent nodal involvement.
Time Frame: From first dose of blinatumomab up to the end of study. Median (min, max) time on study was 188.0 days (19.0, 1512.0).
Population: Full Analysis Set: Included all participants who received blinatumomab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort Ia: Blinatumomab 9/28 µg/Day + Pembrolizumab | Cohort IIa: Blinatumomab 9/28/56 µg/Day + Pembrolizumab | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab
Number analyzed (Participants) | 12 | 10 | 9
months | 4.2 (0.7) [0.7 to 24.1] | 1.9 (0.6) [0.6 to 12.8] | 2.8 (1.4) [1.4 to 6.8]

11. Secondary Outcome: Cohort IIIa Only: Progression Free Survival Using the Lugano Classification
Description: Progression-free survival was calculated as the time from the date of the first dose of blinatumomab until the date of diagnosis of progression of lymphoma using the Lugano 2014 classification, or date of death, whichever was earliest.
  For diagnosis of progression of lymphoma, the progression of radiographic assessment of PET-CT using the Lugano Classification was used. Participants who were alive and did not have progression were censored at the last radiological non-missing evaluable tumor assessment date.
  Progressive disease per the Lugano criteria is a score of 4 or 5 on the 5PS with an increase in intensity of uptake from baseline and/or new FDG-avid foci consistent with lymphoma.
Time Frame: From first dose of blinatumomab up to the end of study. Median (min, max) time on study was 188.0 days (19.0, 1512.0).
Population: Full Analysis Set: Included all participants who received blinatumomab with available post-baseline response per the Lugano classification.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab
Number analyzed (Participants) | 9
months | 4.8 [2.8 to NA] — Upper limit was not estimable due to low number of events.

12. Secondary Outcome: Overall Survival
Description: Overall survival was calculated as the time from the date of first dose of blinatumomab until death due to any cause. Participants who were alive at the analysis date were censored at the date last known to be alive.
Time Frame: From first dose of blinatumomab up to the end of study. Median (min, max) time on study was 188.0 days (19.0, 1512.0).
Population: Full Analysis Set: Included all participants who received blinatumomab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort Ia: Blinatumomab 9/28 µg/Day + Pembrolizumab | Cohort IIa: Blinatumomab 9/28/56 µg/Day + Pembrolizumab | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab
Number analyzed (Participants) | 12 | 10 | 9
months | 9.2 [0.7 to NA] — Upper limit was not estimable due to low number of events. | 7.0 [0.7 to NA] — Upper limit was not estimable due to low number of events. | NA [1.4 to NA] — Median and upper limit were not estimable due to low number of events.

13. Secondary Outcome: Duration of Response for Participants Who Achieved CR/PR Using the Revised Response Cheson Criteria
Description: Duration of response was calculated from the date a response of CR or PR was first achieved until the earliest date of a disease assessment indicating a disease progression or death, whichever occurred first. Participants who did not have a relapse event were censored on their last radiological non-missing evaluable tumor assessment date.
Time Frame: From first dose of blinatumomab up to the end of study. Median (min, max) time on study was 188.0 days (19.0, 1512.0).
Population: Full Analysis Set: Included all participants with a CR or PR during the first 12 weeks of blinatumomab treatment according to the revised response criteria were included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort Ia: Blinatumomab 9/28 µg/Day + Pembrolizumab | Cohort IIa: Blinatumomab 9/28/56 µg/Day + Pembrolizumab | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab
Number analyzed (Participants) | 2 | 3 | 3
months | NA [NA to NA] — Median, lower limit and upper limit were not estimable due to low number of events. | 27.0 [5.5 to NA] — Upper limit was not estimable due to low number of events. | 4.4 [0.9 to NA] — Upper limit was not estimable due to low number of events.

14. Secondary Outcome: Cohort IIIa Only: Duration of Response for Participants Who Achieved CMR/PMR Using the Lugano Classification
Description: The duration of response was calculated from the date a response of CMR or PMR was first achieved until the earliest date of a disease assessment indicating a disease progression using the Lugano classification or death, whichever occurred first.
  Participants who did not have a relapse event were censored on their last radiological non-missing evaluable tumor assessment date.
Time Frame: From first dose of blinatumomab up to the end of study. Median (min, max) time on study was 188.0 days (19.0, 1512.0).
Population: Full Analysis Set: Included all participants with a CMR or PMR during the first 12 weeks of blinatumomab treatment according to the Lugano classification.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab
Number analyzed (Participants) | 1
months | 8.0 [NA to NA] — Lower and upper limit were not estimable due to low number of events.

15. Secondary Outcome: Blinatumomab Steady State Concentration (Css)
Description: Serum blinatumomab concentrations were quantified using a validated enzyme-linked immunosorbent assay (ELISA). The lower limit of quantification (LLOQ) for the assay is 50 pg/mL.
  The Css of serum blinatumomab was summarized as the average of the observed concentrations collected after 24 hours from the start of continuous IV infusion or start of the dose step.
  For calculation of Css at 9 µg/day and 28 µg/day dosing, participants in all cohorts were combined.
Time Frame: Day 2 for 9 µg/day Css (all cohorts), days 10, 15, 22, 29, and 43 for 28 µg/day Css (Cohort Ia), day 10 for 28 µg/day Css (Cohorts IIa and IIIa), and days 19, 26, and 40 for 56 µg/day and 112 µg/day Css (Cohorts IIa and IIIa respectively).
Population: Pharmacokinetic Analysis Set: Included all participants who received any infusion of blinatumomab or pembrolizumab and had at least 1 pharmacokinetic sample collected.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Blinatumomab 9 µg/Day: Participants received blinatumomab administered via a continuous intravenous infusion of 9 µg/day.
- Blinatumomab 28 µg/Day: Participants received blinatumomab administered via a continuous intravenous infusion of 28 µg/day.
- Blinatumomab 56 µg/Day: Participants received blinatumomab administered via a continuous intravenous infusion of 56 µg/day.
- Blinatumomab 112 µg/Day: Participants received blinatumomab administered via a continuous intravenous infusion of 112 µg/day.
Arm/Group | Blinatumomab 9 µg/Day | Blinatumomab 28 µg/Day | Blinatumomab 56 µg/Day | Blinatumomab 112 µg/Day
Number analyzed (Participants) | 27 | 24 | 3 | 2
pg/mL | 280 (215) | 711 (307) | 1380 (478) | 2090 (396)

16. Secondary Outcome: Blinatumomab Clearance
Description: Systemic clearance (CL) was calculated as CL=R0/Css,DN; where R0 is the infusion rate (μg/hr) and Css,DN is the dose normalized average Css.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: liters/hour
Arm/Group | Cohort Ia: Blinatumomab 9/28 µg/Day + Pembrolizumab | Cohort IIa: Blinatumomab 9/28/56 µg/Day + Pembrolizumab | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab
Number analyzed (Participants) | 12 | 9 | 8
liters/hour | 1.84 (0.829) [lower limit 0.829] | 2.06 (0.432) [lower limit 0.432] | 1.76 (0.614) [lower limit 0.614]

17. Secondary Outcome: Pembrolizumab Peak Serum Concentration
Description: Pembrolizumab serum concentrations were quantified using a validated electro-chemiluminescent-based immunoassay with a lower limit of quantification of 25 ng/mL.
  The pembrolizumab pharmacokinetic data from all cohorts were combined for analysis.
Time Frame: Within approximately 30 minutes after the end of the infusion in cycle 1 (study day 15 for Cohort Ia, study day 19 for Cohorts IIa and IIIa) and cycle 8 (study day 162 for Cohort Ia and day 166 for Cohorts IIa and IIIa).
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Blinatumomab + Pembrolizumab: Participants received blinatumomab administered CIVI for 8 weeks followed by a 28-day treatment-free interval. For Cohort Ia, the starting dose was 9 μg/day for the first 7 days and then the dose was increased to 28 μg/day for the remainder of the treatment period. For Cohorts IIa and IIIa, the dose was 9 μg/day for the first 7 days, was escalated to 28 μg/day for next 7 days, then was increased to a maximum of 56 μg/day in Cohort IIa, or to 112μg/day in Cohort IIIa from Day 15. Starting on study day 15 in Cohort Ia, and on study day 19 in Cohorts IIa and IIIa, participants also received 200 mg pembrolizumab administered by IV infusion Q3W until disease progression or for up to 35 cycles.
Arm/Group | Blinatumomab + Pembrolizumab
Number analyzed (Participants) | 21
μg/mL
  Cycle 1 | 52.7 (24.7)
  Cycle 8: number analyzed (Participants) | 5
  Cycle 8 | 124 (27.8)

18. Secondary Outcome: Pembrolizumab Minimum Serum Concentration
Description: Pembrolizumab serum concentrations were quantified using a validated electrochemiluminescent-based immunoassay with a lower limit of quantification of 25 ng/mL.
  The pembrolizumab pharmacokinetic data from all cohorts were combined for analysis.
Time Frame: Pre-dose on pembrolizumab cycles 2, 4, 6, 8, and 12 (Study days 36, 78, 120, 162, and 246, respectively).
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Blinatumomab + Pembrolizumab: Participants received blinatumomab administered CIVI for 8 weeks followed by a 28-day treatment-free interval. For Cohort Ia, the starting dose was 9 μg/day for the first 7 days and then the dose was increased to 28 μg/day for the remainder of the treatment period. For Cohorts IIa and IIIa, the dose was 9 μg/day for the first 7 days, was escalated to 28 μg/day for next 7 days, and then was increased to a maximum of 56 μg/day in Cohort IIa, or to 112μg/day in Cohort IIIa from Day 15. Starting on study day 15 in Cohort Ia, and on study day 19 in Cohorts IIa and IIIa, participants also received 200 mg pembrolizumab administered by IV infusion Q3W until disease progression or for up to 35 cycles.
Arm/Group | Blinatumomab + Pembrolizumab
Number analyzed (Participants) | 16
μg/mL
  Cycle 2 | 13.9 (25.7)
  Cycle 4: number analyzed (Participants) | 11
  Cycle 4 | 34.2 (29.9)
  Cycle 6: number analyzed (Participants) | 9
  Cycle 6 | 50.5 (23.1)
  Cycle 8: number analyzed (Participants) | 6
  Cycle 8 | 62.6 (27.3)
  Cycle 12: number analyzed (Participants) | 3
  Cycle 12 | 53.2 (15.7)

19. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as any untoward medical occurrence in a clinical trial participant that started after the initiation of blinatumomab.
  All TEAEs were graded using NCI CTCAE Version 4.0:
  * Grade 2: Moderate
  * Grade 3: Severe or medically significant but not immediately life-threatening.
Time Frame: From first dose of blinatumomab to minimum of 30 days after last dose of blinatumomab or pembrolizumab (whichever was later) or end of study: median (min, max) duration was 22.7 (1.0, 85.8) days.
Population: Safety Analysis Set: Included all participants who received blinatumomab.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort Ia: Blinatumomab 9/28 µg/Day + Pembrolizumab | Cohort IIa: Blinatumomab 9/28/56 µg/Day + Pembrolizumab | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab
Number analyzed (Participants) | 12 | 10 | 9
Participants
  TEAEs | 12 | 10 | 9
  Grade ≥ 2 TEAEs | 12 | 10 | 9
  Grade ≥ 3 TEAEs | 11 | 9 | 9

ADVERSE EVENTS:
Time Frame: Mortality- From enrollment to end of study: median (min, max) was 188.0 (19.0 ,1512.0) days. TEAEs - From first dose of blinatumomab to minimum of 30 days after last dose blinatumomab/pembrolizumab: median (min, max) was 22.7 (1.0, 85.8) days.
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- Cohort Ia: Blinatumomab 9/28 µg/Day + Pembrolizumab: Participants in Cohort Ia received blinatumomab administered as a CIVI for 8 weeks followed by a 28-day treatment-free interval. Participants with stable disease or better may have received a second 28-day consolidation cycle. The starting dose of each cycle was 9 µg/day for the first 7 days, then 28 µg/day for the remaining days of treatment. Starting on Day 15 participants also received 200 mg pembrolizumab administered by IV infusion Q3W until disease progression or for up to 35 cycles.
- Cohort IIa: Blinatumomab 9/28/56 µg/Day + Pembrolizumab: Participants in Cohort IIa received blinatumomab administered as a continuous intravenous infusion for 8 weeks followed by a 28-day treatment-free interval. Participants with stable disease or better may have received a second 28-day consolidation cycle. The starting dose of each cycle was 9 µg/day for the first 7 days, 28 µg/day for 7 days, then 56 µg/day for the remaining days of treatment. Starting on Day 19 participants also received 200 mg pembrolizumab administered by IV infusion Q3W until disease progression or for up to 35 cycles.
- Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab: Participants in Cohort IIIa received blinatumomab administered as a continuous intravenous infusion for 8 weeks followed by a 28-day treatment-free interval. Participants with stable disease or better may have received a second 28-day consolidation cycle. The starting dose of each cycle was 9 µg/day for the first 7 days, 28 µg/day for 7 days, then 112 µg/day for the remaining days of treatment. Starting on Day 19 participants also received 200 mg pembrolizumab administered by IV infusion Q3W until disease progression or for up to 35 cycles.
Arm/Group | Cohort Ia: Blinatumomab 9/28 µg/Day + Pembrolizumab | Cohort IIa: Blinatumomab 9/28/56 µg/Day + Pembrolizumab | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 6/12 | 7/10 | 4/9
Serious Adverse Events (participants affected / at risk) | 9/12 | 7/10 | 9/9
Other Adverse Events (participants affected / at risk) | 12/12 | 10/10 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort Ia: Blinatumomab 9/28 µg/Day + Pembrolizumab (N=12) | Cohort IIa: Blinatumomab 9/28/56 µg/Day + Pembrolizumab (N=10) | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab (N=9)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Vestibular ataxia (Ear and labyrinth disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 1
Disease progression (General disorders) | 5 | 3 | 1
Performance status decreased (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 1
Bacillus bacteraemia (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Staphylococcus test positive (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 6
Apraxia (Nervous system disorders) | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 1
Coordination abnormal (Nervous system disorders) | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 0 | 2
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 1
Neurological symptom (Nervous system disorders) | 0 | 0 | 1
Neurotoxicity (Nervous system disorders) | 0 | 0 | 3
Seizure (Nervous system disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Hallucinations, mixed (Psychiatric disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Malignant ascites (Gastrointestinal disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Hypersomnia (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort Ia: Blinatumomab 9/28 µg/Day + Pembrolizumab (N=12) | Cohort IIa: Blinatumomab 9/28/56 µg/Day + Pembrolizumab (N=10) | Cohort IIIa: Blinatumomab 9/28/112 µg/Day + Pembrolizumab (N=9)
Anaemia (Blood and lymphatic system disorders) | 3 | 5 | 3
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 4 | 2 | 2
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 0
Ear swelling (Ear and labyrinth disorders) | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 1 | 0
Eye allergy (Eye disorders) | 1 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 1
Periorbital swelling (Eye disorders) | 0 | 1 | 0
Photophobia (Eye disorders) | 1 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0
Anal erythema (Gastrointestinal disorders) | 0 | 0 | 1
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0
Duodenogastric reflux (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 3 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 2 | 2
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1
Tongue spasm (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 2
Asthenia (General disorders) | 1 | 1 | 1
Catheter site erythema (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Chills (General disorders) | 1 | 2 | 0
Disease progression (General disorders) | 1 | 1 | 0
Face oedema (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 5 | 3 | 1
Generalised oedema (General disorders) | 1 | 0 | 0
Inflammation (General disorders) | 0 | 1 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0
Mass (General disorders) | 1 | 0 | 0
Nodule (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 2 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 1
Pain (General disorders) | 2 | 0 | 3
Peripheral swelling (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 5 | 3 | 5
Swelling face (General disorders) | 0 | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 2 | 1
Hypogammaglobulinaemia (Immune system disorders) | 2 | 0 | 1
Balanitis candida (Infections and infestations) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 1 | 0
Lower respiratory tract infection fungal (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 3 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 3 | 2
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Amylase increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 2 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0
Cortisol decreased (Investigations) | 1 | 0 | 0
Enterococcus test positive (Investigations) | 0 | 0 | 1
Fibrin D dimer increased (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 1
Helicobacter test positive (Investigations) | 0 | 0 | 1
Hepatic enzyme abnormal (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 3 | 3 | 2
Neutrophil count decreased (Investigations) | 1 | 1 | 3
Platelet count decreased (Investigations) | 3 | 3 | 1
Weight decreased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 3 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 3 | 3
Hypouricaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 2
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 6 | 3 | 2
Horner's syndrome (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0
Neurological symptom (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 3
Agitation (Psychiatric disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 2 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Ureteric compression (Renal and urinary disorders) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Central venous catheterisation (Surgical and medical procedures) | 0 | 1 | 0
Ureteral stent insertion (Surgical and medical procedures) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Spontaneous bacterial peritonitis (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Synovial rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Aspartate aminotransferase abnormal (Investigations) | 1 | 0 | 0
Candida test positive (Investigations) | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Superficial vein thrombosis (Vascular disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Based on the results of Part 1, a decision was made not to proceed with Part 2 of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT03340766/Prot_002.pdf
  • Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT03340766/SAP_003.pdf